CLINICAL TRIAL: NCT01021176
Title: A Single Dose Pilot Study to Evaluate the Safety and Dose-Response of Smell to Intranasal Diltiazem
Brief Title: Evaluate a Medication on How Hunger and Appetite Are Influenced by Smell
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Compellis Pharmaceuticals (Unknown)
Responsible Party: Principal Investigator, Frank Greenway, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PBRC 27016
Record Dates: First submitted 2009-11-24; First posted 2009-11-26 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Food Intake
Keywords: Food Intake; Hunger; Lidocaine; Nose; smell
MeSH Terms: conditions — Anosmia | interventions — Diltiazem

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0mg 0 spray (Placebo Comparator): No Diltiazem
  Interventions: Other: Placebo spray
- 2mg 2 Spray (Active Comparator): Staff member will administer an atomizer (device that changes a liquid into a fine spray) that will go into both nostrils. The atomizer will contain diltiazem, RxC Use 2mg/2 spray Diltiazem
  Interventions: Drug: Diltiazem
- 4mg 4 Spray (Active Comparator): Staff member will administer an atomizer (device that changes a liquid into a fine spray) that will go into both nostrils. The atomizer will contain diltiazem, RxC Use 4mg/4 spray Diltiazem
  Interventions: Drug: Diltiazem
- 8mg 8 spray (Active Comparator): Staff member will administer an atomizer (device that changes a liquid into a fine spray) that will go into both nostrils. The atomizer will contain diltiazem, RxC Use 8mg/8 spray Diltiazem
  Interventions: Drug: Diltiazem

INTERVENTIONS:
Other: Placebo spray — 0, 30, 60, 90, 120, 180, and 240 minutes following the nasal spray yet no drug will be administered
  Other Names: Placebo
  Arms: 0mg 0 spray
Drug: Diltiazem — 0, 30, 60, 90, 120, 180, and 240 minutes following the nasal spray Three Dilutions would be 5.5, 6.0 and 6.3 and the fourth at the filp of a coin randomly diluted.
  Other Names: 5.5, 6.0, 6.3 and/or one more randomly
  Arms: 2mg 2 Spray; 4mg 4 Spray; 8mg 8 spray

SUMMARY:
The purpose of this study is to determine whether the blood pressure medication, diltiazem, will temporarily decrease the sense of smell when given in a nasal spray which will then reduce food intake.

DETAILED DESCRIPTION:
You will fast on your first visit. Complete questionnaire about taste and smell to insure you don't have a cold or anything that would interfere with sense of smell. Your nose will be checked. Blood pressure taken, and administer to you a spray with diltiazem 2, 4, 8 mg or a placebo. Your sense of smell will be tested at different time points.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 25 and 40 kg
* Blood pressure in within normal range

Exclusion Criteria:

* Used tobacco products in the past month
* Used a calcium channel blocker medication in the last month
* used nasal sprays in the last month
* have an abnormal sense of smell or abnormalities of the lining in your nose
* female and have irregular menstrual periods
* female and are nursing a baby or pregnant
* female and have had a partial hysterectomy (still have ovaries)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Evidence of blood pressure medication, diltiazem, will temporarily decrease the sense of smell when given in a nasal spray. | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frank L. Greenway, MD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States